CLINICAL TRIAL: NCT06831149
Title: A Phase 2 Trial of Intraoperative Fluorescent Angiography to Decrease Pharyngocutaneous Fistula Rates in Patients Undergoing Hypopharyngeal Reconstruction
Brief Title: Use of SPY Imaging System to Minimize Fistulas After Hypopharyngeal Reconstruction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew Spector (Other)
Responsible Party: Sponsor-Investigator, Matthew Spector, Professor of Otolaryngology - Head and Neck Surgery and Chief of the Head and Neck Surgery and Oncology Division., University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24100162
Record Dates: First submitted 2025-02-13; First posted 2025-02-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Carcinoma; Pharyngocutaneous Fistula
Keywords: squamous cell carcinoma hypopharynx; squamous cell carcinoma larynx; SPY Fluorescence Imaging System
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Prospective, interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients having salvage TL after failure with radiation or chemoradiation (Other): SPY intraoperative fluorescent angiography system to risk stratify patients intraoperatively into low and high risk groups for developing pharyngocutaneous fistula (PCF) postoperatively
  Interventions: Procedure: Removal of pharyngeal mucosa with decreased perfusion will be performed; Device: SPY-PHI; Drug: ICG (Indocyanine Green)

INTERVENTIONS:
Procedure: Removal of pharyngeal mucosa with decreased perfusion will be performed — Surgical removal of underperfused tissue versus nonremoval of tissue
Device: SPY-PHI — SPY Portable Handheld Imaging (SPY-PHI)
Drug: ICG (Indocyanine Green) — ICG will be used in conjunction with the SPY-PHI system for tissue imaging.

SUMMARY:
Investigators performing this research want to look at the use of a special imaging process during a specific throat surgery. Using this imaging may help to lower a common complication that called a pharyngocutaneous fistula (PCF). A PCF is a leak in the tube in the throat that helps with breathing and digesting food.

The imaging is called the SPY Fluorescence System. This system can identify tissue that is not receiving enough blood. The SPY Fluorescence System uses a special dye, called Indocyanine green (ICG) to better see the tissues that are not receiving enough blood. When tissue does not receive enough blood, it can lead to infection. Infection of tissue in this area of the throat can lead to PCF. The imaging takes about 1 minute and is performed in the operating room during surgery.

For this study, the investigators (who are also surgeons) will decide to remove tissue that is identified by the SPY Fluorescence System to have decreased blood flow. They will then continue with the rest of the surgery as usual. The investigators will monitor participants as they recover from surgery to identify any complications that may occur. For this research they are interested in complications during the first month after surgery since this is when PCF usually happens.

Investigators will use information that has been documented in the medical records of participants as well as during in-person physical examinations during inpatient recovery and outpatient clinical visits.

DETAILED DESCRIPTION:
Our prior work has demonstrated the efficacy to predict pharyngocutaneous fistula using Indocyanine green (ICG) angiography. In an observational study of 41 patients who underwent salvage TL with onlay free flap reconstruction, 7 (17%) patients developed PCF. Intraoperative angiography has the ability to measure the blood flow rate (ingress) into the tissues. In patients with ingress <15 (n=25), 24% developed a PCF. In contrast, no PCF was seen in the group with ingress >15. Of note, in patients with ingress <15, there was no intervention performed as this was an observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Prior diagnosis of biopsy-proven squamous cell carcinoma of the larynx or hypopharynx (stage II-IV)
2. Prior treatment with radiation +/- chemotherapy
3. Presence of local recurrence of disease, radiation necrosis or an incompetent larynx
4. 18 years or older. 5. Ability to understand and sign informed consent

Exclusion Criteria:

1. Iodine and Shellfish allergy
2. Contraindication to surgery under general anesthesia
3. Anticipated extended laryngectomy (laryngopharyngectomy or laryngopharyngoesophagectomy) with the need for free tissue transfer to reconstruct the pharyngeal mucosa. This may only be determined at the time of surgery
4. Pregnancy or lactation.
5. Patients residing in prison.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of PCF, within one month post total laryngectomy (TL) | From enrollment through 1 month post surgery
  Incidence of PCF, in participants identified as "high risk", utilizing the SPY Fluorescence Imaging System during total laryngectomy (TL) surgical procedure, within one month post TL. Incidence of PCF will be monitored during post operative, inpatient hospitalization as well as clinical outpatient follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew E Spector, MD, Principal Investigator — University of Pittsburgh/UPMC
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
At the time of creation of the project, the investigators do not envision the need to share IPD with other researchers or other entities. The funding for the project is internal so there is no need to report to an external sponsor.